CLINICAL TRIAL: NCT06241105
Title: A Prospective Phase II Clinical Trial of Lenvatinib in Combination With Toripalimab for Patients With Platinum-Resistant Recurrent Ovarian Cancer
Brief Title: Lenvatinib Plus Toripalimab for Platinum-Resistant Recurrent Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: The Second Affiliated Hospital of Dalian Medical University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Fengzhi Feng, professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K3559
Record Dates: First submitted 2024-01-09; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Recurrent Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: Lenvatinib plus Toripalimab
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenvatinib+Toripalimab (Experimental): 1. Administer 8 mg of Lenvatinib orally, once a day, for continuous usage;
  2. Administer 240mg of Toripalimab via intravenous infusion, first time seven days post-lenvatinib intake, and subsequently every three weeks thereafter.
  Interventions: Drug: Lenvatinib+Toripalimab.

INTERVENTIONS:
Drug: Lenvatinib+Toripalimab. — Adjustment of Medication Dosage: Throughout the course of treatment, adjustments should be made exclusively to the dosage of the drug Lenvatinib.The starting dosage for lenvatinib is 8 mg, administered orally once a day for a period of four weeks. If no adverse reactions are observed, the dosage can be escalated to 12 mg for individuals weighing over 60 kg. However, if the patient experiences intolerable side effects, the dosage should be decreased back to 8 mg.For individuals weighing less than 60 kg, the maximum dosage is 8 mg per day. Should adverse reactions become intolerable, the dosage may be decreased to 4 mg per day.Withdrawal from the study if still intolerable.

SUMMARY:
The investigators propose to initiate a study assessing the efficacy and safety of a lower initial dosage of lenvatinib combined with toripalimab in patients suffering from platinum-resistant recurrent ovarian cancer. The objective of this research is to offer a novel therapeutic approach for patients battling relapsed ovarian cancer with platinum resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 75 years;
2. Platinum-resistant recurrence of epithelial ovarian cancer, fallopian tube cancer, and primary peritoneal cancer.
3. According to the RECIST 1.1 criteria, there should be at least one measurable lesion or a CA 125 level of ≥ 70 IU/L.
4. ECOG 0-2；
5. Liver and Kidney Function: Serum creatinine levels should be ≤ 1.5 times the upper limit of the normal range.AST and ALT levels should be ≤ 2.5 times the upper limit of normal, or ≤ 5 times the upper limit of normal if liver metastases are present;total bilirubin should be ≤ 1.5 times the upper limit of the normal range.
6. Participants of reproductive age must consent to the use of effective contraceptive methods throughout the duration of the study.Women of reproductive age must yield a negative result in serum or urine pregnancy tests.Non-lactating patients.
7. Those who are expected to survive longer than 3 months. Patients were unconscious and volunteered to participate in the study.

Exclusion Criteria:

1. Uncontrollable malignant hypertension;
2. Imaging showed that the tumor invaded important blood vessels;
3. Contraindications to the use of antiangiogenic agents;
4. Contraindications to checkpoint inhibitors;
5. Patients presenting with abdominal fistula, gastrointestinal perforation, and pelvic-abdominal abscess;
6. Simultaneous involvement or engagement in another clinical trial within a one-month period that could potentially influence the outcomes of this study.
7. Known hypersensitivity to study-related drugs or their excipients;
8. Individuals with severe heart, liver, kidney, and other serious concurrent diseases that may pose a threat to life;
9. Patients judged by the investigator to be inappropriate for participation in the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 69 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From the start of treatment to a minimum of 3 years
  This term denotes the duration from the initiation of enrollment to the point of neoplasm progression or death.

SECONDARY OUTCOMES:
Overall Survival (OS) | From the start of treatment to a minimum of 3 years
  Overall Survival refers to the duration from the initiation of enrollment until death, regardless of the cause.For participants who have not succumbed, the data will be censored at the most recent date known for their survival.
Objective Response Rate (ORR) | From the start of treatment to a minimum of 3 years
  The Objective Response Rate (ORR) is defined as the sum of the proportions of complete and partial responses. This is achieved when there is a reduction in the neoplasm volume to a predetermined value, coupled with a decrease in serum CA 125 concentration by more than 50% post-treatment compared to pre-treatment levels, sustained for a minimum duration of 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi f Feng, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided